CLINICAL TRIAL: NCT05533593
Title: Analysis of Risk Factors of Aminoglycines Related Acute Kidney Injury in Hospitalized Patients and Development of Machine Learning Model
Brief Title: Risk Factors and Machine Learning Model for Aminoglycines Related Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xiao Li，MD, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: LCYY-LX-20220102
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Aminoglycoside Toxicity; Acute Kidney Injury
Keywords: Aminoglycosides; Acute kidney injury; Pharmacoepidemiology; Miss diagnosis; Risk factors; Logic regression
MeSH Terms: conditions — Acute Kidney Injury | interventions — Aminoglycosides

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI Group
  Interventions: Drug: Aminoglycoside
- Non-AKI Group
  Interventions: Drug: Aminoglycoside

INTERVENTIONS:
Drug: Aminoglycoside — Inpatients using aminoglycoside

SUMMARY:
Drug-induced acute kidney injury (D-AKI) can occur after treatment with aminoglycosides. Predicting the risk of D-AKI is important for a tailored prevention and palliation strategy. There are currently no studies to construct a model for predicting the risk of D-AKI associated with aminoglycosides. Therefore, the study aimed to develop a model to predict the risk of D-AKI that could be used in clinical practice. Clinical data of inpatients treated with aminoglycosides at the First Affiliated Hospital of Shandong First Medical University from January 2018 to December 2020, were collected. The primary endpoint was D-AKI, defined according to the 2012 Global Outcomes for Kidney Disease Improvement (KDIGO). Patient clinical information, including demographic information, admission and discharge information, disease history, medication information, and laboratory tests, was obtained through an in-hospital electronic medical record system. Independent risk factors associated with D-AKI will be screened by univariate and multifactorial analyses. Covariates with significant differences (P < 0.05) were included in logistic regression models. The models were evaluated by the area under the curve (AUC) of the receiver operating characteristic curve (ROC) obtained by ten-fold cross-validation. Future studies are needed to test the application of this model in clinical practice to determine whether D-AKI in this setting can be predicted and mitigated.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients who used aminoglycosides during hospitalization
* Hospital stay ≥ 48h
* Age ≥18 years
* There are two or more blood creatinine tests during hospitalization

Exclusion Criteria:

* Hospital stay < 48h
* Age <18 years
* Glomerular filtration rate (GFR) < 30ml/min/1.73m2 within 48 hours after admission
* AKI was diagnosed on admission
* Less than two Scr test results during hospitalization
* The Scr values were always lower than 40 μmol/L during hospitalization
* Cases with incomplete medical history information

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were included if received treatment with aminoglycosides and discharged from the hospital between January 1, 2018 and December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The incidence of acute kidney injury in hospitalized patients treated with aminoglycosides | Through study completion，up to half a year.
  To analyze the incidence of acute kidney injury in hospitalized patients after using aminoglycosides and to build a prediction model.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao Li，MD, Jinan, Shandong, China

REFERENCES:
- [Derived] Zhang P, Chen Q, Lao J, Shi J, Cao J, Li X, Huang X. Machine learning modeling for the risk of acute kidney injury in inpatients receiving amikacin and etimicin. Front Pharmacol. 2025 May 22;16:1538074. doi: 10.3389/fphar.2025.1538074. eCollection 2025. PMID 40487395